CLINICAL TRIAL: NCT06470321
Title: Identifying Biomarkers of Stress-induced Neurophysiological Changes and Emotion Regulation Deficits to Predict Relapse During Nicotine Abstinence
Brief Title: Biopsychosocial Predictors of Nicotine Relapse
Acronym: BioNic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Panos Zanos, Assistant Professor of Neuropharmacology, University of Cyprus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101031962; 101031962 (Other Grant/Funding Number: European Commission Marie Skłodowska-Curie)
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Smoking; Smoking Cessation; Nicotine Addiction; Tobacco Smoking Behavior
Keywords: Nicotine; Relapse; Vulnerability; Biomarkers; EEG; HRV; Stress Reactivity
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder; Recurrence

STUDY DESIGN:
Intervention Model Description: Intervention Model: Single Group Assignment This is a single-arm study where all participants will receive the same smoking cessation intervention after completing the initial assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smoking Cessation Intervention (Experimental): Participants receive Flexiquit, an avatar-led computerized smoking cessation program. Flexiquit is a self-delivered app providing: motivational interviewing, psychoeducation on addiction/withdrawal, cognitive-behavioral strategies for cravings, relapse prevention, stress/emotion regulation skills. Delivered over 6 months starting Day 2 after initial assessments. Adherence monitored. Biochemical verification of abstinence at 3 and 6 months post-quit.
  Interventions: Behavioral: Flexiquit Computerized Smoking Cessation Program

INTERVENTIONS:
Behavioral: Flexiquit Computerized Smoking Cessation Program — Flexiquit is an avatar-led, self-directed computerized program delivering evidence-based techniques to assist with smoking cessation. It includes motivational interviewing, psychoeducation on nicotine addiction, cognitive-behavioral strategies for coping with cravings, relapse prevention, and stress/emotion regulation skills training. Participants receive the program over 6 months and their adherence is monitored. The program provides tailored feedback to support abstinence.

SUMMARY:
This study aims to investigate the associations between emotion regulation ability, stress-induced neural activity changes, and susceptibility to relapse in smokers attempting to quit. Participants will undergo assessments of emotion regulation, neural activity via quantitative electroencephalography (qEEG), and stress responses before and during a 24-hour nicotine abstinence period. They will then participate in a computerized smoking cessation intervention, and their abstinence status will be monitored for 6 months.

DETAILED DESCRIPTION:
The study will examine the unique and interactive effects of emotion regulation ability (a trait-like vulnerability factor) and biomarkers of stress responses (emotion regulation and neural activation changes) prior to smoking cessation, on cravings, abstinence adherence, and response to a smoking cessation intervention.

The study will be divided into three main phases:

* Ad libitum nicotine use (Day 1): Participants will smoke as usual. Baseline assessments of emotion regulation (heart rate variability), neural activity (qEEG), stress responses (salivary cortisol), and nicotine craving will be conducted before and after exposure to a stress task.
* Acute 24-hour abstinence (Day 2): Participants will abstain from smoking for 24 hours. Emotion regulation, neural activity, withdrawal symptoms, and cue-induced cravings will be assessed.
* Smoking cessation intervention (Days 3 to 180): Participants will engage in a computerized smoking cessation program. Abstinence will be biochemically verified at 3 and 6 months post-quit. Smoking lapses and time to relapse will also be monitored.

The primary outcomes are maintenance of abstinence, smoking lapses, and time to relapse. Secondary outcomes include changes in emotion regulation, neural activity, stress responses, withdrawal symptoms, and cue-induced cravings.

The study hypothesizes that smokers who fail to maintain long-term abstinence will exhibit enhanced stress-induced high-frequency qEEG oscillations, disrupted connectivity in emotion regulation brain regions, and emotion regulation deficits. It is also hypothesized that the interplay between these measures will predict smoking cessation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Smoking at least 10 cigarettes daily for at least 2 years
* Intention to quit smoking
* Medication-free

Exclusion Criteria:

* Presence of psychiatric or medical treatment
* Pregnancy
* Current unstable medical illness
* Recent (prior 6 months) drug or alcohol use disorder
* Major Depression
* Diagnosis of psychotic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Abstinence | Measured at 3 and 6 month follow-ups
  Defined as biochemically verified (via expired carbon monoxide) continuous abstinence from smoking for the full 6 month period after the quit date
Time to First Smoking Lapse | 6 months
  Defined as the number of days between the quit date and the first smoking lapse (smoking even a puff of a cigarette). Smoking lapses will be monitored continuously via self-report.

SECONDARY OUTCOMES:
Withdrawal Symptoms | Baseline, 24 hours
  Assessed via standardized withdrawal symptom questionnaires at baseline and after 24 hours of abstinence.
Emotion Regulation | Baseline, 24 hours
  Measured via heart rate variability before and after stress exposure at baseline and 24-hour timepoints
Neural Activity | Baseline, 24 hours
  Quantitative EEG spectral power and coherence between brain regions involved in emotion regulation assessed at baseline and after 24-hour abstinence.
Stress Responses | Baseline, 24 hours
  Salivary cortisol levels measured before and after stress exposure at baseline and 24-hour timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Applied Neuroscience, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karekla M, Panayiotou G, Collins BN. Predictors of urge to smoke under stressful conditions: An experimental investigation utilizing the PASAT-C task to induce negative affect in smokers. Psychol Addict Behav. 2017 Nov;31(7):735-743. doi: 10.1037/adb0000309. Epub 2017 Aug 28. PMID 28845999
- [Background] Karekla M, Savvides SN, Gloster A. An Avatar-Led Intervention Promotes Smoking Cessation in Young Adults: A Pilot Randomized Clinical Trial. Ann Behav Med. 2020 Oct 1;54(10):747-760. doi: 10.1093/abm/kaaa013. PMID 32383736